CLINICAL TRIAL: NCT00000346
Title: Cognitive Correlates of Substance Abuse, Part 1
Brief Title: Cognitive Correlates of Substance Abuse - 11
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-3-0010-11; Y01-3-0010-11
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2002-12

CONDITIONS: Amphetamine-Related Disorders
Keywords: amphetamine dependence
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Counseling

INTERVENTIONS:
Behavioral: counseling

SUMMARY:
The purpose of this study is to characterize the cognitive performance of methamphetamine abusers by comparing them with cocaine abusers and normal controls.

ELIGIBILITY:
Inclusion Criteria:

M/F . Meet DSM-IV criteria for cocaine or methamphetamine dependence. Agree to conditions of the study and sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States